CLINICAL TRIAL: NCT05936580
Title: Nuwiq Dosing and Outcomes In the ManagEment of Women/Girls With Haemophilia A Needing FVIII Treatment for Surgery - an International, Open-label, Non-controlled Study (NuDIMENSION)
Brief Title: Nuwiq Dosing and Outcomes In the ManagEment of Women/Girls With Haemophilia A Needing FVIII Treatment for Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENA-23
Record Dates: First submitted 2023-06-08; First posted 2023-07-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nuwiq (Experimental): All patients receiving Nuwiq (recombinant FVIII). Nuwiq will be administered intravenously in accordance with the relevant prescribing information. Treatment will be repeated as necessary every 8-24 hours until adequate wound healing, then - if required - for at least another 7 days to maintain FVIII plasma levels of 30-60 IU/dL.
  Interventions: Drug: Nuwiq

INTERVENTIONS:
Drug: Nuwiq — Nuwiq is a purified B-domain-deleted FVIII glycoprotein synthesised by a genetically engineered human embryonic kidney cell line (HEK 293F).

SUMMARY:
Recombinant factor VIII for the prevention of bleeding in women/girls with haemophilia A undergoing major surgery

DETAILED DESCRIPTION:
Female patients with mild to moderate haemophilia A will often need FVIII concentrates to provide haemostatic cover during major surgery. This prospective, open-label, non-controlled, single-arm, multinational, multicentre study aims to evaluate the overall perioperative haemostatic efficacy of Nuwiq in women/girls over 12 with haemophilia A undergoing major surgery requiring FVIII treatment

ELIGIBILITY:
Inclusion Criteria:

1. Women/girls with haemophilia A (FVIII:C ≥1-<40%) according to medical history. Additionally, women/girls with documented FVIII activity levels between ≥ 40% and 50% may be included if there is a documented history of clinically significant bleeding episodes consistent with haemophilia A; and/or either documented prior treatment with FVIII concentrates or a clinical indication that FVIII treatment would have been appropriate (e.g., use of FVIII from a family member, or treatment with alternative haemostatic agents due to access limitations)
2. At least 12 years of age
3. Scheduled to undergo major surgery* requiring FVIII treatment, including elective and emergency procedures and caesarean section in pregnant women with haemophilia A
4. Freely given written informed consent of the patient, or parent/legal representative where applicable, obtained in accordance with local regulations

Exclusion Criteria:

1. Coagulation disorder other than haemophilia A
2. Present or past FVIII inhibitor (≥0.6 Bethesda units [BU]/mL)
3. Severe liver or kidney disease (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] levels >5 times the upper limit of normal; or creatinine >120 μmol/L)
4. Known hypersensitivity to Nuwiq's active substance or its excipients (sucrose, sodium chloride, calcium chloride dihydrate, arginine hydrochloride, sodium citrate dihydrate, poloxamer 188)
5. Pregnancy, except in participants with a planned caesarean section
6. Already had surgery in this study
7. Current participation in another interventional clinical trial
8. Treatment with any investigational medicinal product (IMP) within 30 days prior to screening visit

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall haemostatic efficacy | During surgery and until completion of wound healing (e.g. removal of sutures, cessation of drainage, etc.) as defined by the investigator, during the study duration of 30 ± 3 days after the day of surgical procedure
  Overall haemostatic efficacy of treatment measured as binary "success" or "failure". The overall perioperative haemostatic efficacy of Nuwiq will be adjudicated by an Independent Data Monitoring Committee (IDMC) and determined using a composite assessment algorithm that considers the surgeon's assessment of intraoperative haemostatic efficacy and the investigator's assessment of postoperative haemostatic efficacy to classify the overall haemostatic efficacy as success or failure.

SECONDARY OUTCOMES:
Intraoperative haemostatic efficacy | During surgery: From first skin incision to last suture
  Assessment of intraoperative haemostatic efficacy of Nuwiq using a 4-point ordinal scale:
  Excellent: Intraoperative blood loss was lower than or equal to the average expected blood loss for the type of procedure performed in a patient with normal haemostasis and of the same sex, age, and stature
  Good: Intraoperative blood loss was higher than the average expected blood loss but lower or equal to the maximal expected blood loss for the type of procedure in a patient with normal haemostasis.
  Moderate: Intraoperative blood loss was higher than the maximum expected blood loss for the type of procedure performed in a patient with normal haemostasis, but haemostasis was controlled.
  None: Haemostasis was uncontrolled, necessitating a change in the clotting factor replacement regimen.
Postoperative haemostatic efficacy | During surgery and until completion of wound healing (e.g. removal of sutures, cessation of drainage, etc.) as defined by the investigator, during the study duration of 30 ± 3 days after the day of surgical procedure
  Assessment of postoperative haemostatic efficacy of Nuwiq using a 4-point ordinal scale:
  Excellent: No postoperative bleeding or oozing that was not due to complications of surgery. All postoperative bleeding (due to complications of surgery) was controlled with Nuwiq as anticipated for the type of procedure.
  Good: No postoperative bleeding or oozing that was not due to complications of surgery. Control of postoperative bleeding due to complications of surgery required increased dosing with Nuwiq or additional injections not originally anticipated for the type of procedure.
  Moderate: Some postoperative bleeding and oozing that was not due to complications of surgery. Control of postoperative bleeding required increased dosing with Nuwiq or additional injections not originally anticipated for the type of procedure.
  None: Extensive uncontrolled postoperative bleeding and oozing.
Allogenic blood products | During surgery and until completion of wound healing (e.g. removal of sutures, cessation of drainage, etc.) as defined by the investigator, during the study duration of 30 ± 3 days after the day of surgical procedure
  Use of allogeneic blood products (red blood cells, platelets, and other blood products)
FVIII plasma levels | ≤30 minutes before and 15-30 minutes after Nuwiq injection
  Perioperative plasma levels
Perioperative haemostatic efficacy per WFH criteria | ≤30 minutes before and 15-30 minutes after Nuwiq injection
  Assessed using 4-point scale recommended by WFH:
  Excellent: Intra- and post-operative blood loss similar to non-haemophilic patient. No extra doses of FVIII/bypassing agents needed Good: Intra- and/or post-operative blood loss slightly increased over expectation for non-haemophilic patient, but judged to be clinically insignificant. No extra doses of FVIII/bypassing agents needed Fair: Intra- and/or post-operative blood loss increased over expectation for the non-haemophilic patient, and additional treatment needed. Extra dose of FVIII/bypassing agents needed, or increased blood component of anticipated transfusion requirement Poor: Significant intra- and/or post-operative blood loss substantially increased over expectation for non-haemophilic patient, requires intervention not explained by medical issue other than haemophilia. Unexpected hypotension, unexpected transfer to ICU due to bleeding, substantially increased blood component of the anticipated transfusion requirement
Adverse events | From start of first Nuwiq injection to 30 ±3 days following the surgical procedure
  Incidence of adverse events recorded during the full study period
Thrombotic events | From start of first Nuwiq injection to 30 ±3 days following the surgical procedure
  Incidence of thrombotic events during the study
FVIII inhibitor formation | From start of first Nuwiq injection to 30 ±3 days following the surgical procedure
  Incidence of FVIII inhibitor formation

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Oldenburg, Principal Investigator — Experimental Haematology and Transfusion Medicine, University Clinic Bonn
Locations (15):
- UT Health San Antonio, San Antonio, Texas, United States
- Helsinki University Hospital,Coagulation Disorder Unit, Helsinki, Finland
- France (2):
  - Avenue de la République, Chambray-lès-Tours
  - CHU de Nantes Hôtel-Dieu, Nantes
- Germany (3):
  - Universitätsklinikum Bonn,Institut für Experimentelle Haematologie und Transfusionsmedizin, Bonn
  - Gerinnungszentrum Rhein-Ruhr, Duisburg
  - Universitätsklinikum Hamburg Eppendorf,II. Medizinische Klinik und Poliklinik, Hamburg
- Italy (2):
  - Aziendo Ospedaliera "Puglieze Ciaccio", Catanzaro
  - Policlinico "P. Giaconne", Palermo
- Clinical Center for Serbia, Belgrade, Serbia
- Spain (2):
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Insel Spital Bern, Bern, Switzerland
- St. James's University Hospital, Leeds, United Kingdom
- Centro Hospitalario Pereira Rossell, Montevideo, Uruguay

REFERENCES:
- [Derived] Marquardt N, Langer F, Holstein K, Alvarez Roman MT, Nunez Vazquez R, Miljic P, Drillaud N, Ardillon L, Lehtinen AE, Santoro RC, Napolitano M, Siragusa S, Gidley G, Jansen M, Knaub S, Oldenburg J. Design of an international, phase IV, open-label study of simoctocog alfa in women/girls with hemophilia A undergoing surgery (NuDIMENSION). Ther Adv Hematol. 2024 Dec 1;15:20406207241300040. doi: 10.1177/20406207241300040. eCollection 2024. PMID 39624518